CLINICAL TRIAL: NCT00958113
Title: Autoimmune Thyroid Disease Genetic Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0931
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Hashimoto's Disease; Graves' Disease
MeSH Terms: conditions — Hashimoto Disease; Graves Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autoimmune Thyroid Disease: Patients with Hashimoto's disease or Graves' disease
- Unaffected Population: Population not known to be affected by Hashimoto's Disease or Graves' Disease

SUMMARY:
The hypothesis of this project is that specific genes can be identified that contribute to genetic susceptibility to autoimmune thyroid disease (AITD) in different populations. The specific aim of this project is carry out one or more genomewide association studies (GWAS) to map and ultimately identify genes that confer susceptibility to AITD. AITD consists principally of Hashimoto's Thyroiditis (HT) and Graves' Disease (GD), characterized clinically generally by hypothyroidism and hyperthyroidism, respectively. Both HT and GD are autoimmune diseases characterized by infiltration of the thyroid by T and B cells that are reactive with thyroid antigens and by the production of thyroid autoantibodies (TAB). While there is some evidence that there may be genes specific to either GD or HT, other genes appear to be common to both, and some genes may furthermore be in common to susceptibility to other autoimmune diseases. Genes known to play a role in AITD include HLA, CTLA4, thyroglobulin (TG), THSR, and CD40, PTPN2, and PTPN22, several of which are also involved in susceptibility to other autoimmune diseases. All of these genes interact in a complex manner that has yet to be understood. Furthermore, it seems clear that relatively few of the genes involved in susceptibility to AITD have thus far been discovered.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of abnormal thyroid function (hypo or hyperthyroidism) due to autoimmune thyroid disease

Exclusion Criteria:

* Lack of documentation of abnormal thyroid function or clear evidence of autoimmune etiology

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in Endocrinology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Map and identify genes that confer susceptibility to Autoimmune Thyroid Disease (AITD) | Approximately one year after all samples are collected
  SNP genotypes (allele frequencies, genotype frequencies) will be compared in cases versus controls.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Spritz, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States